CLINICAL TRIAL: NCT01164111
Title: Preoperative Resistance Training in Patients Scheduled for Total Hip Arthroplasty - a Prospective Randomized Study in Patients With Osteoarthritis
Brief Title: Preoperative Resistance Training in Patients Scheduled for Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Andreas Ebbe Bording Hermann, MD, University of Southern Denmark
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: H-4-2010-034
Record Dates: First submitted 2010-07-12; First posted 2010-07-16 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-10

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; hip arthroplasty; resistance training; preoperative training
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Preoperative resistance training (Experimental): preoperative resistance training: Duration 8 weeks. Intensity: 3 sets of 80 % of 1 repetition max (1 RM) in each exercise. Frequency: 2 times/week
  Interventions: Other: Preoperative resistance training
- Control (No Intervention): Standard preoperative track.: No training intervention. Standard preoperative information.

INTERVENTIONS:
Other: Preoperative resistance training — preoperative resistance training: Duration 8 weeks. Intensity: 3 sets of 80 % of 1 repetition max (1 RM) in each exercise (stated as 8-10 repetitions of the exercise). Frequency: 2 times/week. The patient follows a special training program consisting of exercises with knee and hip extension. Training intensity is followed in a personalized log-book for each patient. Sessions are conducted in small teams closely supervised by specially trained physiotherapists.
  Arms: Preoperative resistance training

SUMMARY:
Purpose:

The purpose of this study is to determine the effect of pre operative resistance training on subjects scheduled for total hip arthroplasty due to primary osteoarthritis.

Background:

Decreasing performance with age due to age related muscle loss is well known. Resistance training in elderly has shown significant effect in regaining both muscle force and function.

It has been shown that a chronic condition with limitations in function as seen in osteoarthritis of the hip decreases both muscle performance and size.

Studies of resistance training of the hip related muscle groups in the early postoperative period after total hip arthroplasty have shown significant effect on muscle force and function.

Few studies have investigated preoperative intervention, all with lighter types of training such as water pool training.

The effect of preoperative resistance training on subjects with primal osteoarthritis of the hip is yet to be described.

Study hypothesis:

Preoperative resistance training will significant improve outcomes on both primal and secondary effect parameters pre surgery and at 1 year followup.

DETAILED DESCRIPTION:
BACKGROUND:

Osteoarthritis of the hip is a common condition among elderly. In Denmark 8000 people underwent operation with total hip arthroplasty in 2007, due to osteoarthritis (Danish Register of hip arthroplasty 2007)).

The number of hip arthroplasties has been doubled the last decade mostly due to an increase in the age group 70-79 years (Danish Register of Hip Arthroplasty 2007). The population of elderly has been increased by to the demographic changes (Danish Statistics). A larger need for treatment could be expected in the future due to this development.

The indications of surgery is pain, reduced function and impaired quality of life related to the hip.

Osteoarthritis is divided into two groups: Primary osteoarthritis and secondary osteoarthritis. The cause of primary osteoarthritis is largely unknown. There is a certain amount of genetic predisposition (Felson et al. 1998), the condition is more common among women and the risk of osteoarthritis is larger with higher body weight (Felson et al. 1988) (Anderson et al. 1988).

Secondary osteoarthritis is seen in rheumatoid arthritis, other types of arthritis and due to morphological conditions in the hip like dysplasia (Jacobsen et al 2005).

Aging is followed by loss of muscle mass -a process accentuated in the late senium (Kyle et al 2001). Loss of muscle mass is related to loss of functions in daily living (Kyle et al 2001)(Jannsen et al 2002).

Conditions with impact on daily living, such as osteoarthritis, is likely to accentuate this process even further. It has been shown that unilateral osteoarthritis of the hip is correlated with a reduction in muscle force, muscle size (cross sectional area) and level of neuromuscular activation (Suetta et al 2007), (Suetta et al 2004).

LOSS OF MUSCLE MASS -AN IMPORTANT FACTOR IN PHYSICAL FUNCTION AND TRAINING IN ELDERLY:

The loss of muscle mass is considered one of the most important factors in loss of function and mobility during aging (Volpi et al 2007).

The loss of lean muscle mass (LLM) is substantial during adult life. In young adults LLM contributes with 50 % to the total body mass (Short et al 2000). Studies have shown a 12-14 % loss of LMM and muscle strength pr decade after the age of 40 (Nair et al 1995), (Roth et al 2000), (Porter et al 1995), (Young et al 1985). At the same time muscle fiber types and fiber composition undergo changes along with changes in the hormonal status - both with effect on tissue regeneration (Lexell et al 1995), (Verdijk et al 2007), (Abbasi et al 1993), (Sattler et al 2009).

RESISTANCE TRAINING IN ELDERLY:

Among healthy elderly resistance training (RT) has significant effect on muscle strength (concentric force - 1 repetition max (1RM), maximum isometric force), physical function and body composition (DEXA scan, ultra sound).

In RT studies the training intensity was typically 80% of 1RM (Sillanpää et al 2008), (Sillanpää et al 2009), (Fiatarone et al 1990), (Fiatarone et al 1994), (Hikida et al 2000) 2-3 times a week, in a period of 8-12 weeks (Vandervoort et al 2003).

RESISTANCE TRAINING AND OSTEOARTHRITIS:

There has only been conducted a few studies concerning progressive resistance training in the period around surgery.

Two clinically controlled trials describe progressive resistance training in the post surgery period and only one study describes the effect of genuine progressive resistance training:

Hesse et al (2003) use treadmill training with partly body weight support after hip arthroplasty. They found significant effects on Harris Hip score and manually rated muscle force. Gait speed remained unchanged.

Suetta et al (2004) (2008) use unilateral progressive resistance training of quadriceps muscle groups in a 12 week program post hip arthroplasty. As shown in healthy elderly they find significant effects on outcome measures like physical performance tests (as stair climb, muscular size (computer tomography scan) and max isokinetic knee extension moment.

RESISTANCE TRAINING PRE-SURGERY VERSUS POST-SURGERY

Only few studies describe different training interventions in the preoperative stage in patients with osteoarthritis (D'Lima et al 1996), (Wang et al 2003), (Gilbey et al 2003), (Rodgers et al 1998), (Gill et al 2009). Most of them describe intervention before total knee arthroplasty.

Only 3 studies designed as randomized clinically controlled studies are conducted pre-surgery on patients scheduled for hip arthroplasty (Wang et al 2003), (Gilbey et al 2003), (Gill et al 2009).

All of those with low intensity training like water pool therapy. To our knowledge no studies have described the effect of progressive resistance training as intervention in the pre operative period.

The findings by Suetta et al (2008) of the effect of progressive resistance training post surgery motivates this study of similar intervention in a pre surgery setting.

PURPOSE:

The purpose of this study is:

* To determine the effect of preoperative resistance training on subjects scheduled for total hip arthroplasty due to primary osteoarthritis.
* To determine the effect pre-surgery and post surgery with 1 year follow up.

HYPOTHESIS:

Preoperative resistance training will significant improve outcomes on both primal and secondary effect parameters pre-surgery and at 1 year follow up.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for total hip arthroplasty due to primary osteoarthritis with an age of 50 years or older.
* Patients in the intervention group must participate in 80% of the training as a minimum and more than 2 skipped sessions in a row is not allowed.

Exclusion Criteria:

* Rheumatoid arthritis (RA) or other types of arthritis other than primary osteoarthritis.
* Uremia
* Cancer
* Systemic treatment with glucocorticoid more than 3 months the last 5 years with a daily dose > 5 mg.
* Fracture of the hip (ipsi or contralateral)
* Other fracture of the lower extremities the last year
* Other condition with reduced function (ex polio seq.)
* Weight above 135 kg

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Hip dysfunction and Osteoarthritis Outcome Score (HOOS function -daily living) | 0 weeks (entrypoint =T0)
  Questionnaire on Hip Dysfunktion.
  Rated questions on:
  * symptoms
  * stiffness
  * pain
  * function - daily living
  * function - sports and recreational activities. The questionnaire is validated (compared to WOMAC) in patients with oateoarthritis in the hip - both pre- and postoperative.
Hip dysfunction and Osteoarthritis Outcome Score (HOOS function -daily) | 8 weeks (T1 pre surgery)
  Questionnaire on Hip Dysfunktion.
  Rated questions on:
  * symptoms
  * stiffness
  * pain
  * function - daily living
  * function - sports and recreational activities. The questionnaire is validated (compared to WOMAC) in patients with oateoarthritis in the hip - both pre- and postoperative.
Hip dysfunction and Osteoarthritis Outcome Score (HOOS function - daily living) | 3 months (T3 -post surgery)
  Questionnaire on Hip Dysfunktion.
  Rated questions on:
  * symptoms
  * stiffness
  * pain
  * function - daily living
  * function - sports and recreational activities. The questionnaire is validated (compared to WOMAC) in patients with oateoarthritis in the hip - both pre- and postoperative.
Hip dysfunction and Osteoarthritis Outcome Score (HOOS function - daily living) | 6 months (T4 - postsurgery)
  Questionnaire on Hip Dysfunktion.
  Rated questions on:
  * symptoms
  * stiffness
  * pain
  * function - daily living
  * function - sports and recreational activities. The questionnaire is validated (compared to WOMAC) in patients with oateoarthritis in the hip - both pre- and postoperative.
Hip dysfunction and Osteoarthritis Outcome Score (HOOS function - daily living) | 9 months (T5 -post surgery)
  Questionnaire on Hip Dysfunktion.
  Rated questions on:
  * symptoms
  * stiffness
  * pain
  * function - daily living
  * function - sports and recreational activities. The questionnaire is validated (compared to WOMAC) in patients with oateoarthritis in the hip - both pre- and postoperative
Hip dysfunction and Osteoarthritis Outcome Score (HOOS function - daily living) | 12 months (endpoint - post surgery)
  Questionnaire on Hip Dysfunktion.
  Rated questions on:
  * symptoms
  * stiffness
  * pain
  * function - daily living
  * function - sports and recreational activities. The questionnaire is validated (compared to WOMAC) in patients with oateoarthritis in the hip - both pre- and postoperative

SECONDARY OUTCOMES:
Muscle Power | 0 weeks (pre surgery)
  Bi-articular measurement of mucle power of leg (knee + hip) extension. Explosive muscle power and power-to-weight ratio of the subject measured by the Nottingham Power rig.
Muscle strength | 0 weeks (pre surgery)
  Monoarticular measurement of muscle strength. Knee extension and Hip extension respectively. Muscle power measured by isometric force and rate of force development. Measurements on a secured bench specially build for the purpose.
Functional scores | 0 weeks (pre surgery)
  Functional scores:
  Stair climb test: 10 steps up/down. Gait velocity test: 20 meters walk: normal speed, high speed. Chair sit-to-stand
Body composition: Dual Energy X-ray Absorptiometry scan(DEXA scan) | 0 weeks (pre surgery
  DEXA:
  Whole body and regional scan to estimate body composition (fat/fat free mass)+ bone density (BMD).
Activity score: Metabolic equivalent score (MET- score) | 0 weeks (pre surgery)
  The MET score estimates the metabolic equivalent from an activity questionnaire.
Muscle Power | 8 weeks (pre surgery)
  Bi-articular measurement of mucle power of leg (knee + hip) extension. Explosive muscle power and power-to-weight ratio of the subject measured by the Nottingham Power rig.
Muscle Power | 3 months (post surgery)
  Bi-articular measurement of mucle power of leg (knee + hip) extension. Explosive muscle power and power-to-weight ratio of the subject measured by the Nottingham Power rig.
Muscle Power | 12 months (post surgery)
  Bi-articular measurement of mucle power of leg (knee + hip) extension. Explosive muscle power and power-to-weight ratio of the subject measured by the Nottingham Power rig.
Muscle strength | 8 weeks (pre surgery)
  Monoarticular measurement of muscle strength. Knee extension and Hip extension respectively. Muscle power measured by isometric force and rate of force development. Measurements on a secured bench specially build for the purpose.
Muscle strength | 3 months (post surgery)
  Monoarticular measurement of muscle power. Knee extension and Hip extension respectively. Muscle power measured by isometric force and rate of force development. Measurements on a secured bench specially build for the purpose.
Muscle strength | 12 months (post surgery)
  Monoarticular measurement of muscle strenth. Knee extension and Hip extension respectively. Muscle power measured by isometric force and rate of force development. Measurements on a secured bench specially build for the purpose.
Functional scores | 8 weeks (pre surgery)
  Stair climb test: 10 steps up/down. Gait velocity test: 20 meters walk: normal speed, high speed. Chair sit-to-stand
Functional scores | 3 months (post surgery)
  Stair climb test: 10 steps up/down. Gait velocity test: 20 meters walk: normal speed, high speed. Chair sit-to-stand
Functional scores | 12 months (post surgery)
  Stair climb test: 10 steps up/down. Gait velocity test: 20 meters walk: normal speed, high speed. Chair sit-to-stand
Body composition: Dual Energy X-ray Absorptiometry scan (DEXA scan) | 8 weeks (pre surgery)
  Whole body and regional scan to estimate body composition (fat/fat free mass)+ bone density (BMD).
Body composition: Dual Energy X-ray Absorptiometry scan (DEXA scan) | 3 months (post surgery)
  Whole body and regional scan to estimate body composition (fat/fat free mass)+ bone density (BMD).
Body composition: Dual Energy X-ray Absorptiometry scan (DEXA scan) | 12 months (post surgery)
  Whole body and regional scan to estimate body composition (fat/fat free mass)+ bone density (BMD).
Activity score: Metabolic equivalent score (MET score) | 8 weeks (pre surgery)
  The MET score estimates the metabolic equivalent from an activity questionnaire
Activity score: Metabolic equivalent score (MET score) | 3 months (post surgery)
  The MET score estimates the metabolic equivalent from an activity questionnaire
Activity score: Metabolic equivalent score (MET score) | 6 months (post surgery)
  The MET score estimates the metabolic equivalent from an activity questionnaire
Activity score: Metabolic equivalent score (MET score) | 9 months (post surgery)
  The MET score estimates the metabolic equivalent from an activity questionnaire
Activity score: Metabolic equivalent score (MET score) | 12 months (post surgery)
  The MET score estimates the metabolic equivalent from an activity questionnaire
Hip dysfunction and Osteoarthritis Outcome Score (HOOS symptoms) | 0 weeks presurgery
  Questionnaire on Hip Dysfunktion.
Hip dysfunction and Osteoarthritis Outcome Score (HOOS symptoms, pain, sports &recreation, hip related quality of life) | 8 weeks presurgery
  Questionnaire on Hip Dysfunktion.
Hip dysfunction and Osteoarthritis Outcome Score (HOOS symptoms, pain, sports &recreation, hip related quality of life) | 3 months post surgery
  Questionnaire on Hip Dysfunktion.
Hip dysfunction and Osteoarthritis Outcome Score (HOOS symptoms, pain, sports &recreation, hip related quality of life) | 6 monts post surgery
  Questionnaire on Hip Dysfunktion.
Hip dysfunction and Osteoarthritis Outcome Score (HOOS symptoms, pain, sports &recreation, hip related quality of life) | 9 months post surgery
  Questionnaire on Hip Dysfunktion.
Hip dysfunction and Osteoarthritis Outcome Score (HOOS symptoms, pain, sports &recreation, hip related quality of life) | 12 monts post surgery
  Questionnaire on Hip Dysfunktion.

CONTACTS AND LOCATIONS:
Overall Officials: Andreas EB Hermann, MD, Principal Investigator — University of Southern Denmark
Locations (1):
- Ortopædkirurgisk Afdeling T Herlev Hospital, Herlev, Denmark

REFERENCES:
- [Background] Dansk Hoftealloplastikregister(register of danish hip arthroplasty). Year report 2007
- [Background] Danmarks statistik. www.statistikbanken.dk
- [Background] Felson DT, Couropmitree NN, Chaisson CE, Hannan MT, Zhang Y, McAlindon TE, LaValley M, Levy D, Myers RH. Evidence for a Mendelian gene in a segregation analysis of generalized radiographic osteoarthritis: the Framingham Study. Arthritis Rheum. 1998 Jun;41(6):1064-71. doi: 10.1002/1529-0131(199806)41:63.0.CO;2-K. PMID 9627016
- [Background] Felson DT, Anderson JJ, Naimark A, Walker AM, Meenan RF. Obesity and knee osteoarthritis. The Framingham Study. Ann Intern Med. 1988 Jul 1;109(1):18-24. doi: 10.7326/0003-4819-109-1-18. PMID 3377350
- [Background] Anderson JJ, Felson DT. Factors associated with osteoarthritis of the knee in the first national Health and Nutrition Examination Survey (HANES I). Evidence for an association with overweight, race, and physical demands of work. Am J Epidemiol. 1988 Jul;128(1):179-89. doi: 10.1093/oxfordjournals.aje.a114939. PMID 3381825
- [Background] Jacobsen S, Sonne-Holm S, Soballe K, Gebuhr P, Lund B. Hip dysplasia and osteoarthrosis: a survey of 4151 subjects from the Osteoarthrosis Substudy of the Copenhagen City Heart Study. Acta Orthop. 2005 Apr;76(2):149-58. doi: 10.1080/00016470510030517. PMID 16097538
- [Background] Kyle UG, Genton L, Hans D, Karsegard VL, Michel JP, Slosman DO, Pichard C. Total body mass, fat mass, fat-free mass, and skeletal muscle in older people: cross-sectional differences in 60-year-old persons. J Am Geriatr Soc. 2001 Dec;49(12):1633-40. doi: 10.1046/j.1532-5415.2001.t01-1-49272.x. PMID 11843996
- [Background] Janssen I, Heymsfield SB, Ross R. Low relative skeletal muscle mass (sarcopenia) in older persons is associated with functional impairment and physical disability. J Am Geriatr Soc. 2002 May;50(5):889-96. doi: 10.1046/j.1532-5415.2002.50216.x. PMID 12028177
- [Background] Suetta C, Aagaard P, Magnusson SP, Andersen LL, Sipila S, Rosted A, Jakobsen AK, Duus B, Kjaer M. Muscle size, neuromuscular activation, and rapid force characteristics in elderly men and women: effects of unilateral long-term disuse due to hip-osteoarthritis. J Appl Physiol (1985). 2007 Mar;102(3):942-8. doi: 10.1152/japplphysiol.00067.2006. Epub 2006 Nov 22. PMID 17122381
- [Background] Suetta C, Aagaard P, Rosted A, Jakobsen AK, Duus B, Kjaer M, Magnusson SP. Training-induced changes in muscle CSA, muscle strength, EMG, and rate of force development in elderly subjects after long-term unilateral disuse. J Appl Physiol (1985). 2004 Nov;97(5):1954-61. doi: 10.1152/japplphysiol.01307.2003. Epub 2004 Jul 9. PMID 15247162
- [Background] Volpi E, Nazemi R, Fujita S. Muscle tissue changes with aging. Curr Opin Clin Nutr Metab Care. 2004 Jul;7(4):405-10. doi: 10.1097/01.mco.0000134362.76653.b2. PMID 15192443
- [Background] Short KR, Nair KS. The effect of age on protein metabolism. Curr Opin Clin Nutr Metab Care. 2000 Jan;3(1):39-44. doi: 10.1097/00075197-200001000-00007. PMID 10642082
- [Background] Nair KS. Muscle protein turnover: methodological issues and the effect of aging. J Gerontol A Biol Sci Med Sci. 1995 Nov;50 Spec No:107-12. doi: 10.1093/gerona/50a.special_issue.107. PMID 7493201
- [Background] Roth SM, Ferrell RF, Hurley BF. Strength training for the prevention and treatment of sarcopenia. J Nutr Health Aging. 2000;4(3):143-55. PMID 10936901
- [Background] Porter MM, Vandervoort AA, Lexell J. Aging of human muscle: structure, function and adaptability. Scand J Med Sci Sports. 1995 Jun;5(3):129-42. doi: 10.1111/j.1600-0838.1995.tb00026.x. PMID 7552755
- [Background] Young A, Stokes M, Crowe M. The size and strength of the quadriceps muscles of old and young men. Clin Physiol. 1985 Apr;5(2):145-54. doi: 10.1111/j.1475-097x.1985.tb00590.x. PMID 3888498
- [Background] Lexell J. Human aging, muscle mass, and fiber type composition. J Gerontol A Biol Sci Med Sci. 1995 Nov;50 Spec No:11-6. doi: 10.1093/gerona/50a.special_issue.11. PMID 7493202
- [Background] Verdijk LB, Koopman R, Schaart G, Meijer K, Savelberg HH, van Loon LJ. Satellite cell content is specifically reduced in type II skeletal muscle fibers in the elderly. Am J Physiol Endocrinol Metab. 2007 Jan;292(1):E151-7. doi: 10.1152/ajpendo.00278.2006. Epub 2006 Aug 22. PMID 16926381
- [Background] Abbasi AA, Drinka PJ, Mattson DE, Rudman D. Low circulating levels of insulin-like growth factors and testosterone in chronically institutionalized elderly men. J Am Geriatr Soc. 1993 Sep;41(9):975-82. doi: 10.1111/j.1532-5415.1993.tb06764.x. PMID 8409184
- [Background] Sattler FR, Castaneda-Sceppa C, Binder EF, Schroeder ET, Wang Y, Bhasin S, Kawakubo M, Stewart Y, Yarasheski KE, Ulloor J, Colletti P, Roubenoff R, Azen SP. Testosterone and growth hormone improve body composition and muscle performance in older men. J Clin Endocrinol Metab. 2009 Jun;94(6):1991-2001. doi: 10.1210/jc.2008-2338. Epub 2009 Mar 17. PMID 19293261
- [Background] Sillanpaa E, Hakkinen A, Nyman K, Mattila M, Cheng S, Karavirta L, Laaksonen DE, Huuhka N, Kraemer WJ, Hakkinen K. Body composition and fitness during strength and/or endurance training in older men. Med Sci Sports Exerc. 2008 May;40(5):950-8. doi: 10.1249/MSS.0b013e318165c854. PMID 18408601
- [Background] Sillanpaa E, Laaksonen DE, Hakkinen A, Karavirta L, Jensen B, Kraemer WJ, Nyman K, Hakkinen K. Body composition, fitness, and metabolic health during strength and endurance training and their combination in middle-aged and older women. Eur J Appl Physiol. 2009 May;106(2):285-96. doi: 10.1007/s00421-009-1013-x. Epub 2009 Mar 6. PMID 19266214
- [Background] Fiatarone MA, Marks EC, Ryan ND, Meredith CN, Lipsitz LA, Evans WJ. High-intensity strength training in nonagenarians. Effects on skeletal muscle. JAMA. 1990 Jun 13;263(22):3029-34. PMID 2342214
- [Background] Fiatarone MA, O'Neill EF, Ryan ND, Clements KM, Solares GR, Nelson ME, Roberts SB, Kehayias JJ, Lipsitz LA, Evans WJ. Exercise training and nutritional supplementation for physical frailty in very elderly people. N Engl J Med. 1994 Jun 23;330(25):1769-75. doi: 10.1056/NEJM199406233302501. PMID 8190152
- [Background] Hikida RS, Staron RS, Hagerman FC, Walsh S, Kaiser E, Shell S, Hervey S. Effects of high-intensity resistance training on untrained older men. II. Muscle fiber characteristics and nucleo-cytoplasmic relationships. J Gerontol A Biol Sci Med Sci. 2000 Jul;55(7):B347-54. doi: 10.1093/gerona/55.7.b347. PMID 10898248
- [Background] Vandervoort AA. Aging of the human neuromuscular system. Muscle Nerve. 2002 Jan;25(1):17-25. doi: 10.1002/mus.1215. PMID 11754180
- [Background] Hesse S, Werner C, Seibel H, von Frankenberg S, Kappel EM, Kirker S, Kading M. Treadmill training with partial body-weight support after total hip arthroplasty: a randomized controlled trial. Arch Phys Med Rehabil. 2003 Dec;84(12):1767-73. doi: 10.1016/s0003-9993(03)00434-9. PMID 14669181
- [Background] Suetta C, Magnusson SP, Rosted A, Aagaard P, Jakobsen AK, Larsen LH, Duus B, Kjaer M. Resistance training in the early postoperative phase reduces hospitalization and leads to muscle hypertrophy in elderly hip surgery patients--a controlled, randomized study. J Am Geriatr Soc. 2004 Dec;52(12):2016-22. doi: 10.1111/j.1532-5415.2004.52557.x. PMID 15571536
- [Background] Suetta C, Andersen JL, Dalgas U, Berget J, Koskinen S, Aagaard P, Magnusson SP, Kjaer M. Resistance training induces qualitative changes in muscle morphology, muscle architecture, and muscle function in elderly postoperative patients. J Appl Physiol (1985). 2008 Jul;105(1):180-6. doi: 10.1152/japplphysiol.01354.2007. Epub 2008 Apr 17. PMID 18420714
- [Background] D'Lima DD, Colwell CW Jr, Morris BA, Hardwick ME, Kozin F. The effect of preoperative exercise on total knee replacement outcomes. Clin Orthop Relat Res. 1996 May;(326):174-82. doi: 10.1097/00003086-199605000-00020. PMID 8620638
- [Background] Wang AW, Gilbey HJ, Ackland TR. Perioperative exercise programs improve early return of ambulatory function after total hip arthroplasty: a randomized, controlled trial. Am J Phys Med Rehabil. 2002 Nov;81(11):801-6. doi: 10.1097/00002060-200211000-00001. PMID 12394990
- [Background] Gilbey HJ, Ackland TR, Wang AW, Morton AR, Trouchet T, Tapper J. Exercise improves early functional recovery after total hip arthroplasty. Clin Orthop Relat Res. 2003 Mar;(408):193-200. doi: 10.1097/00003086-200303000-00025. PMID 12616059
- [Background] Rodgers JA, Garvin KL, Walker CW, Morford D, Urban J, Bedard J. Preoperative physical therapy in primary total knee arthroplasty. J Arthroplasty. 1998 Jun;13(4):414-21. doi: 10.1016/s0883-5403(98)90007-9. PMID 9645522
- [Background] Gill SD, McBurney H, Schulz DL. Land-based versus pool-based exercise for people awaiting joint replacement surgery of the hip or knee: results of a randomized controlled trial. Arch Phys Med Rehabil. 2009 Mar;90(3):388-94. doi: 10.1016/j.apmr.2008.09.561. PMID 19254601
- [Derived] Holsgaard-Larsen A, Hermann A, Zerahn B, Mejdahl S, Overgaard S. Effects of progressive resistance training prior to total HIP arthroplasty - a secondary analysis of a randomized controlled trial. Osteoarthritis Cartilage. 2020 Aug;28(8):1038-1045. doi: 10.1016/j.joca.2020.04.010. Epub 2020 May 4. PMID 32376477
- [Derived] Hermann A, Holsgaard-Larsen A, Zerahn B, Mejdahl S, Overgaard S. Preoperative progressive explosive-type resistance training is feasible and effective in patients with hip osteoarthritis scheduled for total hip arthroplasty--a randomized controlled trial. Osteoarthritis Cartilage. 2016 Jan;24(1):91-8. doi: 10.1016/j.joca.2015.07.030. Epub 2015 Aug 15. PMID 26285180